CLINICAL TRIAL: NCT00904514
Title: Request to Conduct Research for Same Use of Stored Human Samples, Specimens, or Data Collected in a Terminated NCI-IRB Protocol
Brief Title: Study of Previously Collected and Stored Tissue Samples From Patients Previously Enrolled in a Completed National Cancer Institute Clinical Trial
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000573913; NCI-08-C-N013; P07268
Record Dates: First submitted 2009-05-16; First posted 2009-05-19 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2012-02

CONDITIONS: Cancer
Keywords: recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; Waldenström macroglobulinemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; prolymphocytic leukemia; recurrent mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; recurrent colon cancer; stage IV esophageal cancer; recurrent esophageal cancer; recurrent bladder cancer; stage IV bladder cancer; recurrent ovarian epithelial cancer; epithelial mesothelioma; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; recurrent squamous cell carcinoma of the nasopharynx; stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; squamous cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent metastatic squamous neck cancer with occult primary; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; cervical squamous cell carcinoma; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; fallopian tube cancer; primary peritoneal cavity cancer; ovarian carcinosarcoma; Brenner tumor; untreated metastatic squamous neck cancer with occult primary; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer; stage II pancreatic cancer; stage III pancreatic cancer; ovarian mucinous cystadenocarcinoma; stage IV pancreatic cancer; recurrent squamous cell carcinoma of the larynx; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Colonic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Ovarian Epithelial; Salivary Gland Neoplasms; Uterine Cervical Neoplasms; Mesothelioma, Malignant; Squamous Cell Carcinoma of Head and Neck; Fallopian Tube Neoplasms; Brenner Tumor; Congenital Abnormalities | interventions — Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at previously collected and stored tissue samples from patients previously enrolled in a completed National Cancer Institute clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Conduct research for same use of stored human samples, specimens, and data collected from patients previously enrolled in a terminated National Cancer Institute-Institutional Review Board clinical trial.
* Correlate plasma levels and pharmacokinetics with disease burden and presence of antibodies.
* Correlate tumor markers with disease burden.
* Determine the utility of tumor markers for following patients after treatment.

OUTLINE: Stored human samples, specimens, and data collected from patients previously enrolled in a terminated National Cancer Institute-Institutional Review Board clinical trial are analyzed for research studies*. Antibodies are neutralized to allow for correlation of ELISA assays for immunogenicity with neutralization assays, which require cytotoxicity assays. In cytotoxicity assays, fresh malignant cells are isolated from blood, bone marrow, lymph nodes, or other tissues and incubated with recombinant immunotoxins to determine their sensitivity. Soluble CD25 assays are used to analyze known marker for B-cell malignancies, particularly those that are CD25-positive. Other candidate tumor markers include soluble IRTA2, soluble CD22, and soluble mesothelin. Skin biopsies retained by the Clinical Pathology Lab are used to study capillary leak syndrome. Other research studies include HLA typing to correlate immunological parameters with response and the PAX-gene tube to obtain RNA for quantitative PCR, evaluate monoclonal immunoglobulin expression, study minimal residual disease, and characterize immunoglobulin gene usage and somatic mutation. RNA microarrays are used to study resistance to immunotoxins. Samples of blood are used to study mechanisms of hemolytic uremic syndrome (HUS) from anti-CD22 immunotoxins. DNA samples are analyzed for complement and/or Factor H mutations that would make a patient more susceptible to HUS. Samples are also analyzed for levels of immunotoxin in blood, urine, and other tissues and for quantification of tumor markers on malignant cells using flow cytometry assays.

NOTE: *Assays that have significant risk to the patient or to the patient's family, including genetic cancer susceptibility studies, will not be performed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples available from patients previously enrolled in one of the following terminated National Cancer Institute-Institutional Review Board clinical trials:

  * Phase I study of LMB-2: NCI-96-C-0064; NCI-T95-0042
  * Phase I study of BL22: NCI-99-C-0014; NCI-T98-0063
  * Phase I study of LMB-9: NCI-98-C-0078; NCI-T98-0005
  * Phase I study of LMB-7: NCI-94-C-0172
  * Phase I study of bolus SS1P: NCI-03-C-0243
  * Phase I study of continuous infusion SS1P: NCI-01-C-0011

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Analyses of stored human samples, specimens, and data collected from patients previously enrolled in a terminated National Cancer Institute-Institutional Review Board clinical trial
Correlation of plasma levels and pharmacokinetics with disease burden and presence of antibodies
Correlation of tumor markers with disease burden
Utility of tumor markers for following patients after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Principal Investigator — National Cancer Institute (NCI)